CLINICAL TRIAL: NCT00621933
Title: Surveillance of Ocular Surface Flora (SURFACE)
Status: Completed | Type: Observational
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Other Study IDs: MA-Zymar-08-001
Record Dates: First submitted 2008-02-13; First posted 2008-02-22 (Estimated); Results first posted 2012-07-18 (Estimated); Last update posted 2019-04-26 (Actual); Status verified 2019-04

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Culture Swabs of the conjunctiva and eyelids
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All Patients Receiving Cataract Surgery: All Patients Receiving Cataract Surgery

SUMMARY:
Topical fluoroquinolones (FQs) have achieved widespread use in ophthalmology for both the treatment and prophylaxis of ocular infections. The present study is set to determine the bacteria present on the ocular surface in patients at the time of cataract surgery and to assess the rate of resistance of ocular isolates to commonly used topical antibiotics.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled to undergo cataract surgery
* Able to provide written informed consent

Exclusion Criteria:

* NSAID in the eye to be swabbed within the past 30 days
* Topical anesthetic, topical antibiotic or antiseptic, or dilating drops in the eye to the swabbed within the past 7 days
* Over-the-counter artificial tear drops or astringent /redness reliever drops (e.g., Visine®, Clear eyes® in the eye to be swabbed on the day of trial
* History of conjunctivitis or any ocular infection within the past 3 months

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cataract Surgery Patients
Sampling Method: Probability Sample
Enrollment: 399 (Actual)
Dates: Start 2007-12; Primary Completion 2008-10 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- Salt Lake City, Utah, United States

REFERENCES:
- [Background] Olson R, Donnenfeld E, Bucci FA Jr, Price FW Jr, Raizman M, Solomon K, Devgan U, Trattler W, Dell S, Wallace RB, Callegan M, Brown H, McDonnell PJ, Conway T, Schiffman RM, Hollander DA. Methicillin resistance of Staphylococcus species among health care and nonhealth care workers undergoing cataract surgery. Clin Ophthalmol. 2010 Dec 10;4:1505-14. doi: 10.2147/OPTH.S14333. PMID 21191448

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This was a culture swab study at a single time-point. No medications were administered and patients were not followed beyond the initial culture.
Groups:
- All Patients: All patients receiving cataract surgery
Period: Overall Study
Arm/Group | All Patients
Started | 399
Completed | 399
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Patients
Number analyzed (Participants) | 399
Age, Customized [Number; unit: participants]
  < 50 years | 6
  Between 50 and 59 years | 61
  Between 60 and 69 years | 126
  Between 70 and 79 years | 138
  Between 80 and 89 years | 60
  Between 90 and 99 years | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 224
  Male | 175

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Staphylococcus Epidermidis Species Susceptible and Resistant to Oxacillin on the Eyelid
Description: Percentage of staphylococcus epidermidis species susceptible and resistant to oxacillin on the eyelid. The minimum inhibitory concentrations (MIC) of each species were determined and compared to oxacillin MIC breakpoints. MIC is the lowest concentration of an antimicrobial that inhibits the visible growth of a microorganism after incubation. For Staphylococcus epidermidis, the oxacillin MIC breakpoints were <= 0.25 ug/ml (susceptible) and >= 0.50 ug/ml (resistant).
Time Frame: Baseline
Population: ITT population. All patients with cultures performed of the ocular surface.
Measure: Number; unit: Percentage of Species
Arm/Group | All Patients
Number analyzed (Participants) | 399
Percentage of Species
  Percentage of Species Oxacillin-Susceptible | 51
  Percentage of Species Oxacillin-Resistant | 48

2. Primary Outcome: Percentage of Staphylococcus Epidermidis Species Susceptible and Resistant to Oxacillin on the Conjunctiva
Description: Percentage of staphylococcus epidermidis species susceptible and resistant to oxacillin on the conjunctiva . The minimum inhibitory concentrations (MIC) of each species were determined and compared to oxacillin MIC breakpoints. MIC is the lowest concentration of an antimicrobial that inhibits the visible growth of a microorganism after incubation. For Staphylococcus epidermidis, the oxacillin MIC breakpoints were <= 0.25 ug/ml (susceptible) and >= 0.50 ug/ml (resistant).
Time Frame: Baseline
Population: ITT population. All patients with cultures performed of the ocular surface.
Measure: Number; unit: Percentage of Species
Arm/Group | All Patients
Number analyzed (Participants) | 399
Percentage of Species
  Percentage of Species Oxacillin-Susceptible | 52
  Percentage of Species Oxacillin-Resistant | 45

3. Secondary Outcome: Percentage of Staphylococcus Aureus Species Susceptible and Resistant to Oxacillin on the Eyelid
Description: Percentage of staphylococcus aureus species susceptible and resistant to oxacillin on the eyelid. The minimum inhibitory concentrations (MIC) of each species were determined and compared to oxacillin MIC breakpoints. MIC is the lowest concentration of an antimicrobial that inhibits the visible growth of a microorganism after incubation. For Staphylococcus aureus, the oxacillin MIC breakpoints were <= 2 ug/ml (susceptible) and >= 4 ug/ml (resistant).
Time Frame: Baseline
Population: ITT population. All patients with cultures performed of the ocular surface.
Measure: Number; unit: Percentage of Species
Arm/Group | All Patients
Number analyzed (Participants) | 399
Percentage of Species
  Percentage of Species Oxacillin-Susceptible | 59
  Percentage of Species Oxacillin-Resistant | 34

4. Secondary Outcome: Percentage of Staphylococcus Aureus Species Susceptible and Resistant to Oxacillin on the Conjunctiva
Description: Percentage of staphylococcus aureus species susceptible and resistant to oxacillin on the conjunctiva. The minimum inhibitory concentrations (MIC) of each species were determined and compared to oxacillin MIC breakpoints. MIC is the lowest concentration of an antimicrobial that inhibits the visible growth of a microorganism after incubation. For Staphylococcus aureus, the oxacillin MIC breakpoints were <= 2 ug/ml (susceptible) and >= 4 ug/ml (resistant).
Time Frame: Baseline
Population: ITT population. All patients with cultures performed of the ocular surface.
Measure: Number; unit: Percentage of Species
Arm/Group | All Patients
Number analyzed (Participants) | 399
Percentage of Species
  Percentage of Species Oxacillin-Susceptible | 70
  Percentage of Species Oxacillin-Resistant | 21

ADVERSE EVENTS:
Description: Serious adverse events and adverse events were not collected/assessed.
Arm/Group | All Patients
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less